CLINICAL TRIAL: NCT01398852
Title: Long Term Safety and Effectiveness of the VEGA UV-A System for Corneal Collagen Cross-Linking in Eyes With Keratoconus or Post-Refractive Corneal Ectasia
Brief Title: Safety and Effectiveness Study of the VEGA UV-A System for Cross-linking in Eyes With Keratoconus and Ectasia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CXL-003
Record Dates: First submitted 2011-07-11; First posted 2011-07-21 (Estimated); Results first posted 2013-03-04 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Keratoconus and Ectasia
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CXL Treatment (Experimental): All eyes to be treated with riboflavin and UV light
  Interventions: Drug: Riboflavin; Device: VEGA UV-A Illumination System

INTERVENTIONS:
Drug: Riboflavin — Riboflavin is a solution that will be delivered to the treatment area
Device: VEGA UV-A Illumination System — This is a portable electronic device designed to deliver a dose of UV-A light to the treatment area

SUMMARY:
The purpose of this research study is to evaluate the long tern safety and effectiveness of cross-linking in eyes with keratoconus and ectasia.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older
* Diagnosis of Keratoconus or Ectasia
* Central or Inferior steepening on the Pentacam map
* Topography consistent with Keratoconus or Ectasia
* BSCVA 20/20 or worse
* Removal of contact lenses for required period of time
* Signed written informed consent
* Willingness and ability to comply with schedule for follow up visits

Exclusion Criteria

* For Keratoconus, a history of previous corneal surgery
* Corneal pachymentry equal to or greater and 400
* Previous ocular condition in the eyes to be treated that may predispose the eye for future complications
* A history of chemical injury or delayed healing
* Pregnancy
* A known sensitivity to the study medications
* Nystagmus or any other condition that would prevent a steady gaze during treatment or other diagnostic tests
* Presence or history of any other condition or finding that makes the patient unsuitable as a candidate

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Woolfson Eye Institute, Atlanta, Georgia
  - Massachusetts Eye And Ear Infirmary, Boston, Massachusetts
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - Laser and Corneal Surgery Assoc. PC, New York, New York
  - Mt Sinai Hospital, New York, New York
  - Pamel Vision & Laser Group, New York, New York
  - Cleveland Clinic-Cole Eye Institute, Cleveland, Ohio
  - ReVision Advanced Laser Eye Center, Columbus, Ohio
  - OSU Department of Ophthalomogy, Columbus, Ohio
  - Dell Laser Consultants, Austin, Texas
  - Slade and Baker Vision Center, Houston, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period started December 2010 and ended June 2012 at medical clinics throughout the country.
Pre-assignment Details: Enrolled participants were excluded from the clinical trial because they failed to meet one or more the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | CXL Treatment
Started | 372 (Due to termination of the study the exact number of participants enrolled is unknown at this time.)
Completed | 0
Not Completed | 372

BASELINE CHARACTERISTICS:
Arm/Group | CXL Treatment
Number analyzed (Participants) | 372
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — The study was terminated prior to data analysis.
  Between 18 and 65 years | NA — The study was terminated prior to data analysis.
  >=65 years | NA — The study was terminated prior to data analysis.
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — The study was terminated prior to data analysis.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — The study was terminated prior to data analysis.
  Male | NA — The study was terminated prior to data analysis.
Region of Enrollment [Number; unit: participants]
  United States | 372

OUTCOME MEASURES:

1. Primary Outcome: Changes in Corneal Curvature
Time Frame: 24 MO
Population: The CXL-003 study was terminated and data analysis was not done. The sponsor, Topcon Medical Systems, decided to terminate the study for administrative reasons only, and not as a result of any safety issues or concerns relating to the study.
Arm/Group | CXL Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | CXL Treatment
Serious Adverse Events (participants affected / at risk) | 0/372
Other Adverse Events (participants affected / at risk) | 0/372

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All such Confidential Information shall remain the property of Topcon, as applicable, and Institution agrees that neither it nor Principal Investigator nor any of its employees or Sub-Investigators, if any, shall disclose any of the Confidential Information to third parties, without the prior written consent of Topcon.